CLINICAL TRIAL: NCT06222931
Title: Effects of Whole Body Vibration in Different Devices on Bone and Muscle Mass, Physical Performance, Quality of Life and Falls in Postmenopausal Women
Brief Title: Effects of Whole Body Vibration in Different Devices on Bone and Muscle Mass in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual do Norte do Parana (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Raphael Goncalves de Oliveira, Professor, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0002_UENP
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Bone Density; Muscles; Physical Functional Performance; Accidental Falls; Quality of Life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triplanar Vibration (synchronous) (Experimental): Triplanar vibration, performed at 25 Hz and 4 mm peak-to-peak displacement, for 5 minutes each session, three times a week. Participants will be positioned standing, with knees semi-flexed at 30º.
  Interventions: Device: Triplanar vibrating platform
- Side-alternating vibration (Experimental): Vibration with alternating side of the base, performed at 25 Hz and 4 mm peak-to-peak displacement, for 5 minutes each session, three times a week. Participants will be positioned standing, with knees semi-flexed at 30º.
  Interventions: Device: Side-alternating vibrating platform
- False vibration (Sham Comparator): Platform identical to the other two used by the experimental groups, configured at 25 Hz, however, without peak-to-peak displacement. The platform starts the engine and emits an operating sound identical to a vibrating platform in operation, but does not generate any mechanical vibration. Participants will be positioned standing, with knees semi-flexed at 30º and must remain on the equipment for 5 minutes each session, three times a week.
  Interventions: Other: Sham vibration

INTERVENTIONS:
Device: Triplanar vibrating platform — Mechanical vibration emitted by triplanar vibrating platforms
  Arms: Triplanar Vibration (synchronous)
Device: Side-alternating vibrating platform — Mechanical vibration emitted by side-alternating vibrating platforms
  Arms: Side-alternating vibration
Other: Sham vibration — Simulated vibration
  Arms: False vibration

SUMMARY:
Postmenopausal women suffer from a series of negative health factors, such as decreased bone and muscle mass and physical performance, increasing the risk of falls and decreasing quality of life. Therefore, intervention strategies aimed at mitigating these factors are essential. A technique that has been studied and can reverse these factors is whole-body vibration (WBV), however studies present contradictory results and the main confounding factor appears to be related to the type of vibration (synchronous or side-alternating). Therefore, the primary objective of this project is to verify the effects of 12 months of whole-body vibration on different devices on bone mineral density measurements in postmenopausal women. As a secondary objective, the effects on muscle mass, physical performance, quality of life and falls will be verified. 228 postmenopausal women will participate in the study and will be randomized to: triplanar vibration (synchronous); side-alternating vibration; or false vibration. The interventions will last 12 months and will occur three times a week on non-consecutive days. The following assessments will be carried out at baseline, 6-months and 12-months: bone mineral density and muscle mass by DXA equipment, muscle thickness by ultrasound, peak torque of the knee extensor and flexor muscles by an isokinetic dynamometer, hand grip, balance static postural and vertical jump on a force platform, dynamic balance using the Timed Up and Go test, SPPB battery, fear (FES-I) and incidence of falls and quality of life (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Being postmenopausal (without menstruating for at least 12 months);
* Not performing physical exercise systematically for at least 6 months;
* Not needing assistance to carry out daily tasks;
* Do not present serious cognitive problems that make it impossible to understand simple commands;
* Do not have serious dysfunctions or implants in the spine, hips or lower limbs;
* Not have neurological diseases or diseases that affect bone metabolism;
* Do not have vascular diseases, arrhythmia, use a pacemaker, suffer from epilepsy or seizures;
* No diseases/problems that affect the retina;
* Do not present severe labyrinthitis or vertigo;
* Not using medication/supplements to increase bone and/or muscle mass for at least 6 months;
* Have not undergone cancer treatment in the last 5 years.

Exclusion Criteria:

* Withdraw from participating in the study for any reason;
* Present adverse events during interventions that cannot be controlled.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Baseline (pre-intervention), 6-months and 12-months
  Bone mineral density of the lumbar spine, total hip, femoral neck and trochanter assessed by DXA, expressed in g/cm2
Appendicular skeletal muscle mass | Baseline (pre-intervention), 6-months and 12-months
  Appendicular skeletal muscle mass assessed by DXA, expressed in kg/m2

SECONDARY OUTCOMES:
Muscle thickness | Baseline (pre-intervention), 6-months and 12-months
  Thickness of the rectus femoris muscle assessed by ultrasound, expressed in cm
Physical Performance | Baseline (pre-intervention), 6-months and 12-months
  SPPB functional test battery composed of: static balance (feet together, semi-tandem, and full-tandem); gait speed test (4m); and 5-time sit-to-stand. All expressed in seconds.
Dynamic balance | Baseline (pre-intervention), 6-months and 12-months
  Timed Up and Go test: time taken to get up from a chair, walk three meters, return and sit down in the chair.
Hand grip strength | Baseline (pre-intervention), 6-months and 12-months
  Handgrip test using a Jamar hydraulic dynamometer, expressed in kg.
Static postural balance | Baseline (pre-intervention), 6-months and 12-months
  Bipedal and semi-tandem postural balance test on a force platform to verify the antero-posterior displacement speed (cm/s), medio-lateral displacement speed (cm/s) and COP area (cm2).
Muscle power | Baseline (pre-intervention), 6-months and 12-months
  Countermovement vertical jump with hands on waist to identify the power of the lower limbs expressed in watts.
Lower limb muscle strength | Baseline (pre-intervention), 6-months and 12-months
  Peak isokinetic torque (N.m) of the knee extensor and flexor muscles (concentric/concentric) evaluated by an isokinetic dynamometer at angular velocities of 60, 180 and 300º/s.
Fear of falls | Baseline (pre-intervention), 6-months and 12-months
  Fear of falls assessed by the falls efficacy scale-international (FES-I), which generates scores from 16 to 64 points.
Health-related quality of life | Baseline (pre-intervention), 6-months and 12-months
  The SF-36 questionnaire will be used, which generates scores of 0-100 points for eight domains of health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil